CLINICAL TRIAL: NCT07304752
Title: Effect of Probe Material (Metallic vs. Plastic) on Peri-implant Probing: a Randomized Clinical Trial.
Brief Title: Effect of Probe Material on Peri-implant Probing
Acronym: METPLA-PP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Principal Investigator, Octavi Camps-Font, Associate Professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 57/2025
Record Dates: First submitted 2025-11-16; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Peri-implant Health; Peri-implant Mucositis
Keywords: Visual Analogue Scale; Peri-implant probing; Probing depth; Emergency profile; Dental implant

STUDY DESIGN:
Intervention Model Description: All clinical measurements will be performed by a single examiner previously trained and calibrated for peri-implant probing in order to ensure consistency and minimize measurement error.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metallic probe (Active Comparator): Metallic UNC-15 periodontal probe (HuFriedy PCPUNC156)
  Interventions: Device: Metallic UNC-15 periodontal probe
- Plastic probe (Experimental): Plastic UNC-15 periodontal probe (HuFriedy PCVO12PT)
  Interventions: Device: Plastic UNC-15 periodontal probe

INTERVENTIONS:
Device: Metallic UNC-15 periodontal probe — Probing performed at six sites per implant with the prosthesis in place and after prosthesis removal, under standardized force (0.20 N).
  Arms: Metallic probe
Device: Plastic UNC-15 periodontal probe — Probing performed at six sites per implant with the prosthesis in place and after prosthesis removal, under standardized force (0.20 N).
  Arms: Plastic probe

SUMMARY:
Evaluate whether the type of probe (plastic vs. metallic) modifies the accuracy of peri-implant probing in single-unit implants, by comparing the probing depth recorded with the prosthesis in place versus without the prosthesis (ΔPD, mm). Secondarily, explore the influence of prosthetic design and implant position on probing values and on other clinical and radiographic parameters.

DETAILED DESCRIPTION:
Randomized clinical trial with two parallel groups. Eligible patients will be randomized (1:1 ratio) to one of two parallel treatment groups:

Group 1 (Metal probe): Peri-implant probing performed with a UNC-15 metallic periodontal probe (HuFriedy PCPUNC156).

Group 2 (Plastic probe): Peri-implant probing performed with a UNC-15 plastic periodontal probe (HuFriedy PCVO12PT).

Primary objective:

To evaluate whether the type of probe (plastic vs metallic) modifies the accuracy of peri-implant probing in single-unit implants, by comparing the probing depth recorded with the prosthesis in place versus without the prosthesis (ΔPS, mm).

Secondary objectives:

To explore the influence of prosthetic design (e.g., emergence profile, crown contour) and implant position on probing depth values and other clinical/radiographic parameters.

To evaluate patient-reported discomfort during peri-implant probing, recorded using a 100-mm visual analogue scale (VAS).

The study was designed in accordance with the international consensus on Implant Dentistry Core Outcome Set and Measurement (ID-COSM), published in the Journal of Clinical Periodontology in 2023. The protocol includes all applicable mandatory outcome domains recommended by this consensus for implant dentistry clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Presence of at least one single-unit bone-level implant rehabilitated with a screw-retained prosthesis directly connected to the implant (no intermediate abutment)
* Implant in function for at least 1 year after prosthetic loading
* No pathological bone loss on periapical radiograph (distance from the most coronal rough surface of the implant to the bone crest < 3 mm)
* Ability to understand and sign informed consent
* Peri-implant health or mucositis, defined according to the 2017 World Workshop criteria:
* Health: no clinical signs of inflammation, lack of profuse (line or drop) bleeding on probing, no increase in probing depth compared to previous records, and no progressive bone loss beyond initial remodeling (<2 mm). In the absence of previous radiographs, radiographic bone level <3 mm without bleeding and/or suppuration on probing.
* Mucositis: presence of bleeding and/or suppuration on probing, no increase in probing depth compared to previous records, and no bone loss beyond initial remodeling (<2 mm). In the absence of previous radiographs, radiographic bone level <3 mm with bleeding and/or suppuration on probing.

Exclusion Criteria:

* Cement-retained restorations or prostheses that cannot be removed
* Systemic antibiotic or anti-inflammatory treatment within the previous 3 months
* Pregnancy or lactation
* Peri-implant treatment within the previous 3 months
* Participation in another clinical trial within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Difference in probing depth with vs. without prosthesis (ΔPS, mm) | Baseline (single clinical visit)
  Difference in peri-implant probing depth (ΔPS) between plastic and metallic probes, measured by a single calibrated examiner at six sites per implant using a standardized probing force (20-25 g).
  Unit of Measure: millimeters (mm) This primary outcome was defined following the mandatory outcome domains recommended by the international consensus on Implant Dentistry Core Outcome Set and Measurement (ID-COSM), published in the Journal of Clinical Periodontology in 2023.

SECONDARY OUTCOMES:
Patient Discomfort During Probing (VAS, 0-100 mm) | Immediately after probing, at the study visit
  Pain/discomfort reported by the patient immediately after peri-implant probing. Unit of Measure: millimeters (0-100 mm VAS) , where 0 is the minimum pain value and 100 is the maximum pain value.

OTHER OUTCOMES:
Probing Depth (PPD, mm) | Baseline (single clinical visit)
  Depth of peri-implant sulcus measured at six sites per implant using standardized probing force (20-25 g). Unit of Measure: millimeters (mm)
Width of Keratinized Mucosa (KM, mm) | Baseline (single clinical visit)
  Distance from the mucosal margin to the mucogingival junction at the buccal aspect.
  Unit of Measure: millimeters (mm)
Mucosal Margin Position (DIM, mm) | Baseline (single clinical visit)
  Distance from the mucosal margin to a fixed reference point. Unit of Measure: millimeters (mm)
Clinical Attachment Level (CAL, mm) | Baseline (single clinical visit)
  Calculated as the sum of PPD and DIM. Unit of Measure: millimeters (mm)
Modified Plaque Index (0-3 scale) | Baseline (single clinical visit)
  Plaque accumulation assessed according to the Modified Plaque Index (Mombelli et al., 1987). Plaque deposits around each implant will be evaluated using the Modified Plaque Index (Mombelli et al., 1987), which scores the presence of plaque or calculus on a 0-3 scale:
  0 = no plaque detected
  1. = plaque detectable only by running a probe across the marginal surface
  2. = plaque visible to the naked eye
  3. = abundance of soft matter or presence of calculus Unit of Measure: Units on a scale (0-3)
Bleeding and/or Suppuration on Probing (presence/absence) | Baseline (single clinical visit)
  Presence or absence of bleeding and/or suppuration at each implant following the 2017 World Workshop criteria.
  Unit of Measure: Yes/No
Implant Type (categorical) | Baseline (single clinical visit)
  Design/type of implant placed. Unit of Measure: Categorical
Implant Position (categorical) | Baseline (single clinical visit)
  Specifying whether the implant was placed at bone level or tissue level Unit of Measure: Categorical .
Implant-Prosthetic Connection Type (categorical) | Baseline (single clinical visit)
  The type of implant-prosthetic connection will be recorded, categorized as internal or external.
  Unit of Measure: Categorical
Emergence Angle (EA, °) | Baseline (single clinical visit)
  The emergence angle (EA) will be measured on standardized periapical radiographs as the angle formed between: The longitudinal axis of the implant, traced as a straight line through the center of the implant body; and a tangent line to the outer surface of the prosthetic restoration at the point where the crown emerges from the implant platform.
  Unit of Measure: degrees (°)
Emergence Profile (EP) | Baseline (single clinical visit)
  The emergence profile was recorded as a qualitative variable describing the contour of the restoration. Its classification was determined based on the emergence angle (EA): it was considered concave when EA < 30°, and convex when EA ≥ 30°.
  Unit of Measure: Categorical
Connection-Contour Distance (mm) | Baseline (single clinical visit)
  Linear distance between implant-abutment connection and contour of the restoration.
  Unit of Measure: millimeters (mm)
Prosthesis Material (type) | Baseline (single clinical visit)
  Material used for the prosthesis (e.g. zirconia or metal-ceramic). Unit of Measure: Categorical (material type)
Titanium Height (mm) | Baseline (single clinical visit)
  This variable applies only to implants restored with zirconia crowns. The vertical height (mm) of the titanium base (Ti-base) supporting the zirconia restoration will be measured.
  Unit of Measure: millimeters (mm)
Patient Satisfaction With the Procedure (VAS, 0-100 mm) | Immediately after probing, at the study visit
  Overall satisfaction with the probing experience. Unit of Measure: millimeters (0-100 mm VAS) , where 0 is the minimum satisfaction value and 100 is the maximum satisfaction value.
Perceived Difficulty of Oral Hygiene (VAS, 0-100 mm) | Immediately after probing, at the study visit
  Self-reported difficulty performing peri-implant hygiene. Unit of Measure: millimeters (0-100 mm VAS) , where 0 is the minimum difficulty performing peri-implant hygiene value and 100 is the maximum value.
Presence of Adverse Events (yes/no) | Immediately after probing, at the study visit
  Presence/absence of pain, bleeding or excessive discomfort during or after probing. Unit of Measure: Yes/No
Peri-implant Diagnosis (health vs mucositis) | Baseline (single clinical visit)
  Diagnosis established based on combined PPD and BOP/SUP criteria following the 2017 World Workshop.
  Unit of Measure: Categorical (Health / Mucositis)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hospital Odontològic Universitat de Barcelona — http://www.hospitalodontologicub.cat/es

DOCUMENTS (1):
  • Informed Consent Form: Informed consent updated (2025-11-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT07304752/ICF_000.pdf